CLINICAL TRIAL: NCT03690674
Title: Lifestyle Enhancement for ADHD Program
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Pooja Tandon, Assistant Professor, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001046; R21AT010041-01 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-10-01 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: ADHD
Keywords: ADHD; Physical Activity; Behavioral Management Training; Mobile Health
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Enhancement for ADHD Program (Experimental): There is no comparison/control arm.
  Interventions: Behavioral: Lifestyle Enhancement for ADHD Program

INTERVENTIONS:
Behavioral: Lifestyle Enhancement for ADHD Program — The LEAP intervention consists of 3 components: 1) an enhanced 8-week, group-based BMT curriculum, 2) parent and child use of the Garmin daily activity tracker accompanied by personalized goal setting, and 3) parent participation in a private Facebook group to encourage PA goal achievement and promote social support and positive parenting.
  Other Names: LEAP

SUMMARY:
The purpose of this study is to investigate if physical activity (PA) can increase in children with Attention Deficit/Hyperactivity Disorder (ADHD) using a modified behavioral management training (BMT) program.

DETAILED DESCRIPTION:
The purpose of this study is to increase physical activity (PA) in children with ADHD using a novel, family-based intervention that promotes PA within the context of evidence-based behavioral management training (BMT) for parents, enhanced with mobile health (mHealth) behavior change strategies. Our first aim is to test the feasibility and acceptability, of an 8-week, family-based, multi-level intervention (BMT-Health) to promote PA in young children with ADHD. Our second aim is to derive an estimate of the effect size of the intervention on PA.

ELIGIBILITY:
Inclusion Criteria:

* age 5-10 years
* ADHD diagnosis
* CGI-S rating >4 and <7
* Per caregiver report, engage in <60 min/day of MVPA for at least 5 days per week
* One adult caregiver willing to participate in the study and complete baseline/follow-up measures
* Caregiver able to complete forms in English
* Caregiver owns a smart phone or similar Garmin compatible mobile device (e.g. iPod Touch) or willing to borrow iPod from study coordinators during the study period
* Agree to install and share data from the Garmin smart phone app with investigators

Exclusion Criteria:

* younger than 5 years old or older than 10 years old
* do not meet criteria for ADHD diagnosis
* Meet diagnostic criteria for psychiatric co-morbidities including Autism Spectrum Disorder, Depressive Disorder, Mood Disorder, Psychotic Disorder, or Intellectual Disability that could interfere with intervention uptake
* Per caregiver report, engage in >60 min/day of MVPA for at least 5 days per week

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Tandon, MD, Principal Investigator — Seattle Children's Hospital; Erin Gonzalez, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 70 participants consisting of 35 dyads (caregver+child) were initially enrolled in the study. 2 dyads withdrew from the study before the group treatment sessions began.
Groups:
- Caregivers - Lifestyle Enhancement for ADHD Program; Children - Lifestyle Enhancement for ADHD Program: There is no comparison/control arm.
  Lifestyle Enhancement for ADHD Program: The LEAP intervention consists of 3 components: 1) an enhanced 8-week, group-based BMT curriculum, 2) parent and child use of the Garmin daily activity tracker accompanied by personalized goal setting, and 3) parent participation in a private Facebook group to encourage PA goal achievement and promote social support and positive parenting.
Period: Overall Study
Arm/Group | Caregivers - Lifestyle Enhancement for ADHD Program | Children - Lifestyle Enhancement for ADHD Program
Started | 35 | 35
Completed | 32 | 32
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Population Description is based on the number of parents that began treatment group. 35 were initially enrolled (provided consent), but 2 withdrew before treatment groups began.
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 7.6 [5 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA)
Description: Measured by accelerometer worn by participating children
Time Frame: Baseline (measured prior to week 1 of Treatment Group) and week 9
Population: Only child participants wore the accelerometer. Number analyzed at post reflects participants who withdrew from study and/or did not complete this measurement.
Measure: Mean (Standard Deviation); unit: Moderate-Vigorous Minutes per day
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 34
Moderate-Vigorous Minutes per day
  Baseline (prior to week 1) MVPA | 53.1 (27.7)
  Week 9 MVPA: number analyzed (Participants) | 26
  Week 9 MVPA | 51.8 (24.4)

2. Primary Outcome: Garmin Wear Time
Description: The length of time (in days) each participant wore the Garmin device as a measure of feasibility
Time Frame: Weeks 1 - 9
Population: 66 participants (33 dyads) who wore the Garmin devices.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 66
Days | 49.18 (14.96)

3. Primary Outcome: Number of Facebook Posts
Description: The amount of contribution to the Facebook page (comments, likes, etc) by each participant is a measure of feasibility
Time Frame: Weeks 1 - 9
Population: 33 caregivers (children were not part of the Facebook groups). 2 dyads dropped out of the study after consent and before group started.
Measure: Mean (Standard Deviation); unit: Facebook Posts
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 33
Facebook Posts | 7.91 (18.92)

4. Primary Outcome: Number of Caregivers With Attendance at the Focus Group
Description: Attendance will be taken at the focus group as a measure of study acceptability
Time Frame: Week 9
Population: 33 dyads were still enrolled and participating at this timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 33
Participants | 29

5. Secondary Outcome: Stop Signal Reaction Time (SSRT) Task Score
Description: Measure of executive function completed by the child. Score is time in ms for participant to respond. Lower score is better.
Time Frame: Baseline to week 9
Population: 28 participant children completed this task.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 28
milliseconds
  Pre | 240.4285714 (59.77019483)
  Post | 244.8214286 (69.76258871)

6. Secondary Outcome: Digit Span (DS) Task - Total Score
Description: Measure of executive function completed by the child. Digit Span Task. Minimum score: 0; Maximum score: 54. Higher score is better outcome.
Time Frame: Baseline to week 9
Population: 29 children completed this assessment at both pre and post timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 29
score on a scale
  Pre | 9.9 (3.177)
  Post | 10.31 (2.753)

7. Secondary Outcome: Finger Windows (FW) Task
Description: Measure of executive function completed by the child
Time Frame: Change between baseline and week 9
Population: This task was not utilized during the study due to study team decision due to time consideration and burden on participants.
Arm/Group | Caregivers - Lifestyle Enhancement for ADHD Program | Children - Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Behavior Rating Inventory of Executive Function (BRIEF)
Description: Measure of executive function completed by the parent. Parent rates whether the child displays each behavior never, sometimes, or often. Global Executive Composite Score: Minimum 35; Maximum 90. Higher score indicates better outcome.
Time Frame: Change between baseline and week 9
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 30
T-Score
  Pre | 71.7 (8.69859)
  Post | 68.4 (8.00259)

9. Secondary Outcome: Impairment Rating Scale (IRS)
Description: Measure of functional impairment completed by the parent. The rating scale measures from 0 to 7, where 0 equals no problem and 7 equals extreme problem. Outcome provided as mean of total raw score. Minimum: 0; Maximum: 100. Higher number indicates higher impairment.
Time Frame: Change between baseline and week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 29
score on a scale
  Pre | 72.2414 (18.13374)
  Post | 64.7586 (18.10417)

10. Secondary Outcome: Alabama Parenting Questionnaire (APQ)
Description: Measure of parenting completed by the parent. The responses are on a 1-5 scale, 1 equals never and 5 equals always. Outcome provided as total raw score. Minimum: 9; Maximum: 45.Higher number indicates better outcome.
Time Frame: Change between baseline and week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 30
score on a scale
  Pre | 23.3 (2.48)
  Post | 22.6 (2.24)

11. Secondary Outcome: Health Behaviors Survey
Description: Measure of physical activity, sleep, media use, medication use and complementary/alternative medicine use. Measure reported is the number of Caregivers responding 'yes' to item.
Time Frame: Baseline and week 9
Population: 29 participants that completed measure at both timepoints.
Measure: Number; unit: participants
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 29
participants
  HBS Item - Needs 1:1 supervision (Pre) | 13
  HBS item - Needs 1:1 supervision - (POST) | 4
  HBS Item - Doesn't do well in a group - PRE | 7
  HBS Item - Doesn't do well in a group - POST | 4

12. Secondary Outcome: Child's Sleep Habits Questionnaire (Pre-school and School-aged Children)
Description: The Child's Sleep Habits Questionnaire (pre-school and school-aged children) is a measure of sleep problems completed by the parent. The parent rates each behavior based on their frequency: 'Usually' if something occurs 5 or more times in a week, 'Sometimes' if it occurs 2-4 times in a week, or 'rarely' if something occurs never or 1 times during a week. Parents can also indicate whether or not a sleep habit is a problem by choosing Yes, No, or Not applicable. Total score provided is the sum of all 33 items. Item units are on a scale of 1 -3 points. The Total score range is 33 - 99. The higher the number, the more sleep problems are indicated for the child.
Time Frame: Baseline and week 9
Population: 24 participants that completed measure at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 24
units on a scale
  Pre | 47 (9.371557339)
  Post | 44 (7.541191233)

13. Secondary Outcome: Conners-3 Questionnaire
Description: Measure of ADHD symptoms reported by the parent. The scale ranges from 0 to 3 with 0 equaling not true at all and 3 equaling very much true. The Conners t-score range from 0 - 100. The higher the number, the worse the outcome.
Time Frame: Change between baseline and week 9
Population: 28 participants that completed measure at both timepoints.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 28
Score on a scale
  Connors Inattention - PRE | 78.71 (11.346)
  Connors Inattention - POST | 75.75 (9.721)
  Connors - Hyperactivity/Impulsivity - PRE | 74.89 (12.968)
  Connors - Hyperactivity/Impulsivity - POST | 71.68 (11.898)
  Connors Aggression/Defiance - PRE | 69.21 (16.601)
  Connors Aggression/Defiance - POST | 63.21 (14.444)

14. Secondary Outcome: Teacher Vanderbilt
Description: Pre and Post measures of ADHD symptoms reported by the teacher. The measure items' scale ranges from 0 to 3, with 0 equaling never and 3 equaling very often. The Inattention outcome measure reported is the average number of items (symptoms) in the Inattention Sub-scale of the Vanderbilt that teachers rated their students as 2 or higher on the 0-3 scale. There are 9 items in the Inattention sub-scale, and the range of Inattention Symptoms reported by the teacher is 0-9. The Hyperactive/Impulsive outcome measure reported is the average number of items (symptoms) in the Hyperactive/Impulsive Sub-scale of the Vanderbilt that teachers rated their students as 2 or higher on the 0-3 scale. There are 9 items in the Hyperactive/Impulsive sub-scale, and the range of Hyperactive/Impulsive Symptoms reported by the teacher is 0-9.The higher the number, the more symptoms teachers are reporting.
Time Frame: Baseline and week 9
Population: 33 teachers that reported according to their experience with participant in their class.
Measure: Mean (Standard Deviation); unit: symptoms
Arm/Group | Lifestyle Enhancement for ADHD Program
Number analyzed (Participants) | 33
symptoms
  Vanderbilt Inattention - teacher-report - PRE | 4.91 (3.263)
  Vanderbilt Inattention - teacher-report - POST | 3.61 (2.989)
  Vanderbilt Hyperactive/Impulsive - teacher-report - PRE | 3.67 (3.266)
  Vanderbilt Hyperactive/Impulsive - teacher-report - POST | 2.64 (2.988)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 8 weeks of treatment group. Participants were not monitored/assessed for adverse events outside of the treatment group timeframe.
Arm/Group | Caregivers - Lifestyle Enhancement for ADHD Program | Children - Lifestyle Enhancement for ADHD Program
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 1/35 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregivers - Lifestyle Enhancement for ADHD Program (N=35) | Children - Lifestyle Enhancement for ADHD Program (N=35)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Mother received a concussion due to accident unrelated to study participation. She missed a group session and had a self-reported decline in physical activity due to her accident.
Stomach Flu (Gastrointestinal disorders) | 0 (0) | 2 (2) — 2 children were reported per parents of having contracted the stomach flu. All recovered within 3-4 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT03690674/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03690674/ICF_000.pdf